CLINICAL TRIAL: NCT03356600
Title: The Prospective,Single Arm, Exploratory Clinical Trial of Apatinib Plus Radiotherapy for Patients With Brain Metastases From Non-Small-cell Lung Cancer
Brief Title: Apatinib Plus Radiotherapy for Patients With Brain Metastases From Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanxi Province Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-SXZL 7
Record Dates: First submitted 2017-11-01; First posted 2017-11-29 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Brain Metastases
Keywords: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — apatinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib plus radiotherapy (Experimental): Apatinib:
  Within 1 week before radiotherapy, the dose of Apatinib were 500mg/daily .During radiotherapy,the dose of Apatinib were 250mg/daily.
  After radiotherapy, if the subject did not have a level 3 or above adverse reaction, investigators consider increasing doses to 500mg.
  Radiotherapy:
  The subjects with 1 to 4 metastases receive stereotactic radiosurgery or stereotactic radiation therapy ,and the subjects with more than 4 metastases receive stereotactic radiosurgery plus whole-brain radiation therapy.
  Interventions: Combination Product: Apatinib plus radiotherapy

INTERVENTIONS:
Combination Product: Apatinib plus radiotherapy — Apatinib:
  Within 1 week before radiotherapy, the dose of Apatinib were 500mg/daily .During radiotherapy,the dose of Apatinib were 250mg/daily.
  After radiotherapy, if the subject did not have a level 3 or above adverse reaction, investigators consider increasing doses to 500mg.
  Radiotherapy:
  The subjects with 1 to 4 metastases receive stereotactic radiosurgery or stereotactic radiation therapy ,and the subjects with more than 4 metastases receive stereotactic radiosurgery plus whole-brain radiation therapy

SUMMARY:
To observe the effectiveness and safety of apatinib combined with radiotherapy for brain metastasis from non-small cell lung cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old, males or females;.
2. According to pathological and histological，the subjects were diagnosed with wild-type non-small-cell lung cancer patients from brain metastasis examinations;
3. Subjects failed first-line standard chemotherapy ;
4. Subjects expected survival of more than 3 months;
5. Eastern Cooperative Oncology Group performance status :0-2 points;
6. The main organ function is normal, that is to meet the following standards:(1) Blood routine examination meets the following standards

   a. Hemoglobin ≥90 g/L；b. Absolute Neutrophil Count≥1.5×10^9/L； c. Platelet ≥80×10^9/L； (2)Blood biochemistry examination meets the following standards

   a.Total Bilirubin <1.5 times the upper normal limit；b.Glutamic transaminase <2.5 times the upper normal limit, glutamic-oxalacetic transaminase <2.5 times the upper normal limit， For patients with liver metastasis ,the Glutamic transaminase and glutamic-oxalacetic transaminase index is less than 5 times the upper normal limit c.Serum Cr was less than 1.25 times the upper normal limit
7. Women of reproductive age must undergo urine tests to eliminate the possibility of pregnancy.During the period of treatment and within 8 weeks after the treatment, the subjects voluntarily adopted appropriate methods of contraception .
8. Subjects volunteered to participate in this study and signed informed consent

Exclusion Criteria:

1. Patients with meningeal metastasis;
2. Patients with intracranial stroke;
3. Previous toxicity associated with chemotherapy and / or radiotherapy persisted;
4. Radiological evidence indicates the presence of an empty or necrotic tumor;
5. Radiological evidence indicates the presence of a central tumor invading large blood vessels;
6. Patients need to be treated with anticoagulants or antiplatelet drugs;
7. The subjects with abnormal coagulation function and bleeding tendency (INR>1.5×ULN、APTT>1.5×ULN);during the past 6 months, the subjects experienced severe thrombosis or clinically related severe bleeding events;In the past 3 months, clinically significant hemoptysis occurred;the subjects had inherited bleeding or thrombosis tendency;
8. Subjects with high blood pressure and whose blood pressure can not be reduced to normal range by antihypertensive drugs;
9. Other investigators believe that patients are not eligible for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The intracranial disease progression free survival time | tumor assesment every 8 weeks,up to 24 months
  To observe the intracranial disease progression free survival time of apatinib combined with radiotherapy for brain metastasis from non-small cell lung cancer patients

SECONDARY OUTCOMES:
Progression free survival time | evaluated in 24 months since the treatment began
  Baseline to measured date of progression or death from any cause
Overall survival | the first day of treatment to death or last survival confirm date ,up to 24 months
  Baseline to measured date of death from any cause
Disease control rate | tumor assesment every 8 weeks,up to 24 months
  Baseline to measured progressive disease
Objective response rate | tumor assesment every 8 weeks,up to 24 months
  Baseline to measured stable disease
Dosage changes of dexamethasone | Dosage changes of dexamethasone every 8 weeks,up to 24 months
  To observe the change of the dosage of dexamethasone before and after treatment
Volume change rate of cerebral edema | Volume change rate of cerebral edema every 8 weeks,up to 24 months
  To observe the change of volume change rate of cerebral edema
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | To observe the safety of therapeutic schedule every 8 weeks,up to 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Cognitive function screening ：Mini-mental state examination (MMSE) | Volume change rate of cerebral edema every 8 weeks,up to 24 months
  The Mini-mental state examination checklist includes 30 problems. Answer the correct question, get 1 points, answer wrong or answer not know, get 0 points, the scale of the total score is 0-30. If the score is 27-30 points, cognitive function is normal; if the score is less than 27, there is cognitive dysfunction. If the score is 21-26 points, there is a mild cognitive impairment. If the score is 10-20 points, there is moderate cognitive impairment. If the score is 0-9 points, there is severe cognitive impairment.
Executive function testing：trail marking test（TMT） | Volume change rate of cerebral edema every 8 weeks,up to 24 months
  The TMT, parts A and B, assesses psychomotor speed and executive function.The A part of the TMT test defined the time range of 0-180 seconds, and the greater the value was, the lower function; the B part of the TMT test defined the time range of 0-300 seconds, and the greater the value, the lower function.
Language function detection ：Hopkins verbal learning test-revised（HVLT-R） | these neurocognitive function tests assesment every 8 weeks,up to 24 months
  The COWA tests verbal fluency and executive function.Within 1 minutes, the subjects say how many words contain one word or within the specified category, each acceptable word counts 1 points, and the repeated words are scored without repetition. The higher the score, the better the function.
Verbal learning and memory:Hopkins verbal learning test-revised（HVLT-R） | these neurocognitive function tests assesment every 8 weeks,up to 24 months
  The HVLT-R assesses aspects of verbal learning and memory, including immediate recall, delayed recall, and delayed recognition.In the HVLT-R test, the range of learning score and delayed recall score was 0-12 points, and the greater the score, the better the function.